CLINICAL TRIAL: NCT00199498
Title: Right Apical Versus Septal Pacing Trial
Acronym: RASP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Raymond Yee, Dr.Raymond Yee MD FRCPC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-04-399; HSREB # 10880 (Other: UWO Ethics)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Heart Block; Heart Failure
Keywords: Permanent Pacemaker Implantation- Lead Position
MeSH Terms: conditions — Heart Block; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septal RV lead placement (Experimental): patient randomized to Septal RV lead placement
  Interventions: Device: Septal RV lead placement
- Apical RV lead placement (Active Comparator): patient randomized to Apical RV lead placement (current standard placement)
  Interventions: Device: Apical RV lead placement

INTERVENTIONS:
Device: Apical RV lead placement — RV lead implanted ( according to randomization )at the apex
  Arms: Apical RV lead placement
Device: Septal RV lead placement — RV lead is implanted (according to randomization), on septum
  Arms: Septal RV lead placement

SUMMARY:
The purpose of this study is to examine whether RV (right ventricular)septal pacing has any effect on LV ( left ventricular) function than RV apical pacing in patients who require ventricular pacing.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effect of RV pacing site on LV systolic function as measured by LVEF (left ventricular ejection fraction).

Secondary objectives of this trial include:

1. to compare the effect of RVSeptal(RVS) versus RVApical(RVA)pacing on other indices of systolic and diastolic LV function
2. to compare the rate of heart failure-related hospitalization between RVS versus RVA pacing
3. to compare new-onset atrial fibrillation and stroke rates between RVS versus RVA pacing
4. to assess the effect of RVA versus RVS pacing on quality of life and functional capacity
5. to compare the rate of successful pacemaker lead implantation, complications and chronic electrical performance of RVS versus RVA pacing

ELIGIBILITY:
Inclusion Criteria:

1. a)Fixed (third degree) AV block b) Atrial Fibrillation with average Ventricular rate on ECG </= 40bpm or mean heart rate on Holter monitor </= 60bpm c) Sinus node Dysfunction with PR interval >/= 300msec d) Paroxysmal, persistent or permanent AF undergoing AV node , AV node/HIS ablation e) 2°AV Block with ≥3:1 block
2. the subject is 18 years of age or older
3. the subject has provided written consent -

Exclusion Criteria:

1. Pre-existing permanent cardiac pacemaker or ICD (defibrillator)
2. Presence of Hypertrophic Obstructive Cardiomyopathy
3. Recent cardiac surgery (</= 30 days)
4. Recent myocardial infarction (</= 30 days)
5. Presence of mechanical prosthetic tricuspid valve
6. Patient inability or unwillingness to comply with study protocol and required study visit schedule
7. Concomitant research study whose protocol would conflict or affect the outcome of this study
8. Patient not expected to survive for the duration of the study follow-up due to co-morbid medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
LV ejection fraction measured by radionuclide ventriculography (RVG). | 2 weeks, 24 months and 36 months

SECONDARY OUTCOMES:
Left ventricular diastolic and systolic function indices 2-D echocardiogram/Doppler (ECHO/DOPP). | 36 months
All cause mortality. | 36 months
Non-fatal thromboembolic events including stroke. | 36 months
Heart failure hospitalization or intravenous drug therapy in an outpatient heart failure clinic. | 36 months
Occurrence of new-onset atrial fibrillation or progression to permanent atrial fibrillation. | 36 months
Symptoms and quality of life scores (DUke Activity Status Index, short form (SF)-12 scores. | 2 weeks, 24 and 36 months
NYHA class using SAS survey, 6 minute hall walk distance. | 2 weeks, 24 and 36 months
lead-related complications such as lead dislodgement, myocardial perforation, lead integrity failure, high pacing threshold | 2 weeks, 24 and 36 months
total implant procedure and fluoroscopy time | Implant

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Yee, MD FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada